CLINICAL TRIAL: NCT02421692
Title: Improving Physical Function in Skilled Nursing Facility Residents
Acronym: SNF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14-2388
Record Dates: First submitted 2015-03-13; First posted 2015-04-21 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Physical Deconditioning

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Usual Care (No Intervention): SNF rehabilitation therapists provide all patients with usual standard of care.
- Progressive Rehabilitation (Experimental): SNF rehabilitation therapists have been trained on principles of progressive rehabilitation strategies and will implement to all eligible patients as new standard of care.
  Interventions: Other: Progressive Rehabilitation

INTERVENTIONS:
Other: Progressive Rehabilitation — Progressive, high-intensity strengthening and functional interventions to facilitate independence with functional activities.
  Arms: Progressive Rehabilitation

SUMMARY:
Each year Medicare spends approximately $31.3 billion on 2.4 million skilled nursing facility (SNF) episodes of care. SNFs rely on interdisciplinary approaches to patient care to maximize rehabilitation potential for return to prior level of function and reduce the risk of adverse events in older adults. However despite a substantial increase in spending on SNF services and minimal change in complexity of the caseload, 68% of patients are below their pre-hospitalization level of function at discharge, 25% return to the community, and 18% are hospitalized. This may be partially explained by current SNF approaches to patient care which foster inactivity and participation in low intensity rehabilitation interventions (preliminary data). Both inactivity and low-intensity interventions may perpetuate further functional decline or impede maximal recovery. The serious implication of risk with functional decline is exemplified by studies which have shown declines in physical function can increase the risk of being re-hospitalized six-fold and may infer other long term effects such as increased risk for mortality, morbidity, and institutionalization. Muscle weakness, reduced cardiorespiratory reserve, and neuromuscular deficits have been attributed to this acute decline in function. However current rehabilitation strategies in SNFs do not promote adequate dose and mode of interventions to induce beneficial systemic adaptations, perhaps due to the lack of evidence on effective rehabilitation protocols for this medically-complex population. Therefore, the investigators have designed an rehabilitation program, which uniquely integrates principles of physiologic tissue overload with strengthening and functional interventions for greater gains in physical function. Data will be collected on the first cohort of patients who cycle through a SNF during Stage 1, in which usual care occurs (5 months). Then, staff training on progressive rehabilitation interventions will occur over 2 months. Finally, data will be collected on a second cohort of patients who cycle through a SNF during Stage 2, in which progressive rehabilitation is implemented by SNF staff (5 months). Given the high turnover of patients in SNFs (average length of stay ~21 days), 2 different cohorts of patients will be studied and the analysis will consist of independent 2-sample t-tests. During Stage 1 and 2, measures of physical function will be assessed on all eligible patients at admission and discharge from SNF. Therapists will be assessed on adherence to the protocol through documentation audits and use of on-site observational checklist. Acceptability of the intervention by the patients will be assessed by a patient satisfaction survey. Any adverse events will be obtained from the medical record and documented. The discharge location of all patients will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Adults older ≥55 years of age who are admitted to a skilled nursing facility following hospitalization
2. Qualify to receive at least physical therapy services.

Exclusion Criteria:

1. Patients with primary diagnoses related to neurological disorders will be excluded as patient needs require more of a motor-control approach versus the proposed high-intensity approach. Such patient populations include:

   1. Parkinson's Disease
   2. Traumatic Brain Injury
   3. Recent Cerebral Vascular Accident
   4. Alzheimer's
2. Patients on hospice care will be excluded as the approach is based on palliative principles. Other patients to be excluded will include those with conditions where strength training is contraindicated (as indicated by the American College of Sports Medicine Guidelines for Exercise Testing and Prescription):

   1. Recent unstable fractures
   2. Advanced congestive heart failure (ejection fracture <30%)
   3. Bone metastasis sites
   4. Tumors in strengthening target areas
   5. Acute illness
   6. Recent myocardial infarction (within 3-6 weeks)
   7. Weight bearing restrictions on graft or fracture sites
   8. Exposed tendon or muscle
   9. Absence of pedal pulses
   10. Presence of a fistula
   11. Platelet levels <50,000/µL.
3. Additional exclusions assessed prior to randomization include a score of less than 21 on the Mini-Mental Status Exam.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change from Admission to Discharge (expected average length of stay 21 days)
  Global measure of lower extremity function, which consists of walking speed, chair stands, and balance tests

SECONDARY OUTCOMES:
Gait Speed | Change from Admission to Discharge (expected average length of stay 21 days)
  Time it takes to walk a 4 meter path

OTHER OUTCOMES:
Patient Satisfaction Survey | Discharge (expected average length of stay 21 days)
  8 question survey, scoring each question on a 1-10 scale (1=not at all and 10=extremely)
Therapist Intervention Compliance | Bi-weekly for 5 months during intervention arm
  Audits of therapist documentation and on-site observations with an objective checklist during treatment sessions
Discharge Location | Discharge (expected average length of stay 21 days)
  Record the discharge location of individuals

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, PT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Gardens on Quail, Arvada, Colorado, United States